CLINICAL TRIAL: NCT04671732
Title: Cost-utility Analysis of Fenestrated Aortic Stents Versus Open Surgery for the Treatment of Complex Abdominal Aortic Aneurysms: a Prospective Multicenter Comparative Cohort Study
Brief Title: Cost-utility Analysis of Fenestrated Aortic Stents Versus Open Surgery for the Treatment of Complex Abdominal Aortic Aneurysms
Acronym: ORFEVAR
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200053
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Complex Abdominal Aortic Aneurysm, ie. Juxtarenal or Suprarenal Aortic Aneurysms, Treated by Fenestrated Endovascular Aortic Aneurysm Repair or Open Repair
Keywords: Vascular surgery; Abdominal aortic aneurysm; Juxtarenal aortic aneurysm; Suprarenal aortic aneurysm; Pararenal aortic aneurysm; fenestrated endovascular aortic aneurysm repair; open repair; Cost effectiveness ratio; Cost / utility analysis
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fenestrated endovascular aortic aneurysm repair (FEVAR)
  Interventions: Procedure: Fenestrated endovascular aortic aneurysm repair
- Open repair (OR)
  Interventions: Procedure: open repair of abdominal aortic aneurysm.

INTERVENTIONS:
Procedure: Fenestrated endovascular aortic aneurysm repair — Fenestrated endovascular aortic aneurysm repair consists in excluding a juxtrenal or suprarenal aneurysm by deploying a covered stent (stent graft) in the aorta so as to created sealing zones on both sides of the aneurysm. Since the proximal sealing is located in the visceral segment of the aorta, fenestrations are created to maintain blod flow in renal and visceral arteries. These fenestrations are custom made for each patient. Brindging covered stents are deployed between each fenestration and corresponding target arteries in order to insure sealing of the system.
  Groups: Fenestrated endovascular aortic aneurysm repair (FEVAR)
Procedure: open repair of abdominal aortic aneurysm. — Open repair of abdominal aortic aneurysms consists in cross-clamping the aorta on both sides of the aneurysm and replace the diseased segment by a prosthetic graft.
  Groups: Open repair (OR)

SUMMARY:
Introduction: Complex abdominal aortic aneurysms (CAA) are defined as abdominal aneurysms that are anatomically unsuitable for a standard endovascular repair because of a short infrarenal neck or no infrarenal neck. These CAAA are usually treated either by fenestrated endovascular aortic repair (FEVAR) or open repair (OR). Data comparing these thechniques remain scarce, mainly consisting of systematic reviews based on retrospective studies. Although mid-term and long-term results remain uncertain, FEVAR has gained widespread acceptance in the vascular community. However, this practice is not evidence base. Beyond clinical results, whether FEVAR is cost-effective or not is not demonstrated. A randomized controlled trial comparing FEVAR and OR is unlikely to be conducted since centers have developed specific expertise and practice, and most of surgeons are not keen to randomize patients. Thus, we believe that a prospective comparative multicentric cohort, with a propensity score and minimization of selection, classification and confusion bias is the most realistic way to provide reliable comparative data on cost effectiveness of FEVAR and OR. Overall, 382 patients are expected to be included (159 in each group).

Objective: The objective of this prospective non-randomized comparative multicenter cohort study is to compare the cost effectiveness incremental ratio at 36 months of FEVAR and OR for CAAA.

Method: Patients with CAAA discussed for FEVAR or OR in 37 french vascular centers in during a two years inclusion period constitute the population study. Preoperative and postoperative clinical and imaging data will are collected prospectively in eCRF forms. QOL before and after treatment is assessed by the E5D5L. The follow-up period is three years. The primary outcome is the Incremental cost-utility ratio (cost/QALY) at 36 months. We plan to minimize indication biases by using a proposensity score (proposnsity score maching and Inverse probablility of treatment weighting) based on clinical and anatomic characteristics. Patient at prohibitive risk for OR are excluded. Patient anatomically unsuitable for FEVAR are also excluded .

Conclusion: This study should provided valuable data on cost effectiveness of FEVAR for CAAA. Sub-goup analysis will be also conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of an abdominal aortic aneurysm greater than 50 mm in diameter, anatomically unsuitable for a standard infrarenal stent graft because of an inadequate infrarenal neck and for which a treatment by FEVAR or OR is considered. The AAA can be identified as follows, according to preoperative imaging:

   * Short-neck or juxtarenal aneurysm: if treated by OR, would require an infrarenal proximal aortic suture, regardless of the level of clamping.
   * Suprarenal aneurysm: if treated by OR, would require a suprarenal/supramesenteric/ supraceliac aortic cross clamping, and a proximal bevelled suture and/or a separate revascularization of at least one renal artery.
   * Type IV thoracoabdominal aneurysm: aneurysm extending up to the level of the diaphragm pillars, requiring a supracoeliac clamping with a proximal bevelled suture and/or separate revascularization of at least one renal artery if treated by open surgery.
2. Patients aged 18 and over
3. Patient who expressed a non-opposition to participating in the study.
4. Patient affiliated to the French healyh care system

Exclusion Criteria:

1. Presence of a type I, II, III or V thoracoabdominal aneurysm according to the modified Crawford Classification.
2. Patients for whom an alternative surgical technique is being considered and listes below: laparoscopic aortic repair, hybrid repair, CHIMPS, surgeon modified stent grafting, in situ fenestrations.
3. Patients deemed at prohibitive risk for OR :

   * uncompensated cardiac failure with LVEF <40% (NYHA class III and IV)
   * Coronary revascularization < 1 month
   * Large myocardial ischemia >3 segments not revascularized or not revascularizable
   * Non-revascularized or non-revascularizable unstable angina
   * Non-operable tight aortic stenosis (mean gradient > 40 mmHg, valve area < 1 cm2, peak transvalvular velocity > 4 m/s)
   * Non operable significant mitral shrinkage (area <1.5cm²)
   * FEV1 < 50% of the theoretical value
   * Home oxygen therapy
   * Chronic renal failure with clearance < 30 ml/min
4. presence of a main renal artery less than 4 mm in diameter
5. Special anatomical configurations: horseshoe kidney, pelvic kidney.
6. Lesions of "shaggy" aorta at the visceral segment or at the lower thoracic aorta
7. History of abdominal aortic surgery (open or endovascular)
8. Dissecting, infected, ruptured or painful aneurysm
9. Life expectancy less than 2 years
10. Person under judicial protection
11. Person under tutorship or curatorship
12. Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with complex AAA (juxtarenal AAA, suprarenal AAA and type IV AAA) needing elective surgical repair (diameter < 50 mm) either by FEVAR or OR.
  Patients at prohibitive risk for OR are excluded. Patients anatomically unsuitable for FEVAR are also excluded.
Sampling Method: Probability Sample
Enrollment: 492 (Actual)
Dates: Start 2021-03-14 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
Incremental cost-utility ratio | at 36 months post-intervention
  cost-effectiveness ratio of fenestrated endovascular aortic aneurysm repair (FEVAR) versus Open repair (OR) in the management of complex AAA in real life

SECONDARY OUTCOMES:
Comparison of quality of life after surgery | at 30 days
  Comparison of quality of life after FEVAR and OR Quality of life 1 month after surgery,as assessed by EQ5D3L questionnaire
Comparison of quality of life after surgery | at 36 months)
  Comparison of quality of life after aortic aneurysm repair or open repair Quality of life 36 months after surgery as assessed by EQ5D3L questionnaire

OTHER OUTCOMES:
36 month mortality | at 36 months
  Comparison of overall and aortic-related mortality rates after aortic aneurysm repair or open repair
Intra-hospital Mortality | at 30 days
  Percentage of deaths after surgery
Number of complications 36 months after the intervention Time frame: short term (< 30 days), medium-term (36 months) after the intervention EPF or CO | at 36 months
  Comparison of complication rates after aortic aneurysm repair or open repair
Number of complications 1 month after the intervention Time frame: short term (< 30 days), medium-term (36 months) after the intervention EPF or CO | at 1 month
  Comparison of complication rates after aortic aneurysm repair or open repair
Number of reintervention after FEVAR and OR surgery | at 1 month
  Comparison of reintervention rates after 1 month FEVAR and OR surgery
Number of reintervention | at 36 month
  Comparison of reintervention rates after 36 month aortic aneurysm repair or open repair

CONTACTS AND LOCATIONS:
Overall Officials: Malika Yahmi, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Assistance Publique Hôpitaux de Paris - CHU HENRI MONDOR, Créteil, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No